CLINICAL TRIAL: NCT02289911
Title: Comparison of Two Learning Methods in Focused Assessment With Sonography for Trauma (FAST) Training Among Paramedics
Brief Title: FAST Learning Methods
Acronym: FAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAST/2014/03
Record Dates: First submitted 2014-11-07; First posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Trauma
Keywords: ultrasound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Class (Active Comparator): Traditional learning form
  Interventions: Other: Didactic training in the FAST
- Web (Active Comparator): Didactic training using internet
  Interventions: Other: Didactic training in the FAST

INTERVENTIONS:
Other: Didactic training in the FAST — Participants in the classroom group (class) listened to traditional lectures, while the web group (web) watched narrated lectures online. All participants completed a pre- and post-test, and a second post-test eight weeks later. Both groups underwent hands-on training after the first post-test.

SUMMARY:
Training paramedics in new skills via classroom-based teaching has inherent costs and time constraints. The investigators sought to evaluate whether web-based didactics result in similar knowledge improvement and retention of FAST (Focused Assessment with Sonography for Trauma) compared with the traditional method.

DETAILED DESCRIPTION:
Paramedics were randomized into a classroom group with traditional lectures and a web group that watched narrated lectures online. All participants completed a pre- and post-test, and a second post-test four weeks later. Both groups underwent hands-on training after the first post-test. A control group completed the two initial tests without didactic intervention.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study emergency medical professionals (paramedics, nurses, physicians)

Exclusion Criteria:

* not meet the above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Knowledge (Mean test scores by didactic group for three consecutive multiple choice tests) | 1 MONTH
  Mean test scores by didactic group for three consecutive multiple choice tests

SECONDARY OUTCOMES:
Self reported satisfaction | 1 MONTH
  Participant satisfaction with training and reported comfort with ultrasound use after training

CONTACTS AND LOCATIONS:
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland